CLINICAL TRIAL: NCT03477357
Title: A Study to Determine the Accuracy of a Non-contact Thermometer in the Perioperative Setting
Brief Title: Accuracy of Non-contact Thermometry
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 214661
Record Dates: First submitted 2017-07-11; First posted 2018-03-26 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Geratherm non Contact thermometer — Temperature taken from subject using non-contact device as per manufacturers instructions

SUMMARY:
Subjects will be admitted to hospital the evening prior, or the morning of surgery, whereupon they will undergo standard admission processes, including pre-operative assessment by the anaesthetist assigned to that list (One of the two study authors). The anaesthetist will then explain the study again, reiterating the potential risks and benefits of the study to the patient themselves, and to the population as a whole. Consent will be sought at this point.

Patients will be transferred to theatre, anaesthetised and operated on as per normal practice. Inclusive of this, in accordance with NICE guidelines, patients will have a nasal or oesophageal Doppler probe inserted to accurately measure core temperature. At this point, patients enrolled in the study will have temperature measurements taken every minute from the oesophageal probe and non-contact thermometers.

If the patients requested it previously, they will be informed of the results of the study at a later date.

Statistics will then be carried out on the data to compare accuracy of the two novel methods to the oesophageal probe.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients undergoing elective gynaecological, vascular or urological surgery at the Royal Sussex County Hospital, and as such will be seen at a pre-operative assessment clinic as part of their normal work up for theatre.

Exclusion Criteria:

- Lacking mental capacity Not speaking English Malignancy in medical history Undergoing open abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be patients undergoing elective gynaecological, vascular or urological surgery at the Royal Sussex County Hospital, and as such will be seen at a pre-operative assesment clinic as part of their normal work up for theatre
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Core body temperature measurement will be taken from 30 patients to compare non-contact infra-red thermometer to oesophageal temperature probes | 12 months
  Bland Altman analysis to compare the readings of 2 methods of temperature measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jack Reid, MBBS, Principal Investigator — BSUH
Locations (1):
- Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be anonymised and analysed later.